CLINICAL TRIAL: NCT03196492
Title: Effect of Injectable Contraceptives on Inflammation, Vaginal Microbiota, and STI/HIV Risk Among Adolescent Girls and Young Women
Brief Title: Vaginal Microbiota, and STI/HIV Risk Among Adolescent Girls and Young Women
Acronym: AIMS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland, College Park (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00126504; 1R01HD092013 (NIH)
Record Dates: First submitted 2017-06-19; First posted 2017-06-22 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No hormone: Half of the cohort (n=40) will have opted to forgo hormonal contraception (HC).
  Interventions: Other: No intervention
- Depo-provera: Half of the cohort (n=40) will have opted to initiate injectable depo-provera (DMPA).

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: No hormone

SUMMARY:
The investigators are doing a study on the bacteria that normally live in the vagina and what effect, if any, Depo-Provera has on the bacteria.

Women 13-24 years of age, who are HIV negative, being seen in a clinic for birth control or sexually transmitted disease (STD) check-up, or have a child and are planning to receive a Depo-Provera shot for contraception or have declined the use of hormonal contraception may join.

DETAILED DESCRIPTION:
The investigators are doing a study on the bacteria that normally live in the vagina and what effect, if any, Depo-Provera has on the bacteria.

Women 13-24 years of age, who are HIV negative, being seen in a clinic for birth control or STD check-up, or have a child and are planning to receive a Depo-Provera shot for contraception or have declined the use of hormonal contraception may join.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-24
* Female sex
* Seeking contraceptive/ STI services OR has had a child OR is legally married
* Has had consensual vaginal sex
* Two years have passed since menses started
* HIV negative by self-report
* Willing to refrain from using douches, washes, or other similar feminine hygiene products. (Tampons are allowed)
* Planning to receive the Depo-Provera shot, -OR- Have regular menstrual cycles with at least 21 - 45 days between menses and plans to use no hormonal birth control.

Exclusion Criteria:

* Any other immunodeficiency (e.g. organ transplant recipient)
* Recently pregnant (within 4 weeks), currently pregnant, or planning to become pregnant within the next 12 months
* Currently breastfeeding
* Hysterectomy or a known genital tract anomaly
* Amenorrhea (except if caused by contraceptive method like the implant)
* Antibiotic or antifungal use within past 30 days

Ages: 13 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy 13-24 Adolescent Girls and Young Women
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Association between lactobacillus-dominant microbiota and sexually transmitted infections (STI) | 6 months
  The investigators will determine if there is an association between lactobacillus-dominant microbiota and STIs. The investigators will report the prevalence of each vaginal community state types (CST) and STIs.

CONTACTS AND LOCATIONS:
Overall Officials: Jenell Coleman Fennell, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No